CLINICAL TRIAL: NCT04408976
Title: Implementation Study With Machine Learning Based Decision Support Software for Treatment of Urinary Tract Infections in General Practice.
Brief Title: Implementation Study With Decision Support Based on Data
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Pacmed BV (Unknown); Zorgverzekeraar CZ (Other); Zorgverzekeraar Zilveren Kruis (Unknown); Zorgverzekeraar Menzis (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Netherlands Instititute for Health Services Research (Other)
Responsible Party: Principal Investigator, Tn Bonten, Assistant Professor, Leiden University Medical Center
Other Study IDs: P1746
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Urinary Tract Infections
Keywords: Machine learning; Clinical Decision Support Systems
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Software practices: Patients with urinary tract infection in practices using the clinical decision support software
- Control practices: Patients with urinary tract infection in practices not using the clinical decision support software

SUMMARY:
This study evaluates the implementation of a machine learning based clinical decision support system for treatment of patients presenting with an urinary tract infection in general practice. The software was developed to support general practitioners in the choice of antibiotic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a urinary tract infection in general practice
* Age > 12 years.

Exclusion Criteria:

* No.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a urinary tract infection diagnosed by the general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 16824 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Non-recurrent UTI | 28 days
  A subsequent period of time after treatment, in which no new UTI treatment was needed

CONTACTS AND LOCATIONS:
Overall Officials: Willem Herter, Study Director — Leiden University Medical Center; Tobias Bonten, Principal Investigator — Leiden University Medical Center
Locations (1):
- Netherlands Institute for Health Services Research, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herter WE, Khuc J, Cina G, Knottnerus BJ, Numans ME, Wiewel MA, Bonten TN, de Bruin DP, van Esch T, Chavannes NH, Verheij RA. Impact of a Machine Learning-Based Decision Support System for Urinary Tract Infections: Prospective Observational Study in 36 Primary Care Practices. JMIR Med Inform. 2022 May 4;10(5):e27795. doi: 10.2196/27795. PMID 35507396